CLINICAL TRIAL: NCT06949033
Title: Neoadjuvant Cadonilimab Combined With Perioperative Oxaliplatin Plus S1 for Diffuse or Mixed Type of Locally Advanced Gastric/Gastroesophageal Junction Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Zuoyi Jiao (Other)
Responsible Party: Sponsor-Investigator, Zuoyi Jiao, Medical Professor, Lanzhou University Second Hospital
Organization: Lanzhou University Second Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LanzhouU2H-2025A-017
Record Dates: First submitted 2025-03-30; First posted 2025-04-29 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-03

CONDITIONS: Gastric Cancer (Including Stomach and Gastroesophageal Junction [GEJ]); Neoadjuvant Therapy; Adjuvant Chemotherapy; pCR Rate; MPR; ORR,OS,PFS
Keywords: gastric cancer; Diffuse or Mixed type; Cadonilimab; Oxaliplatin; S1
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Neoadjuvant cadonilimab combined with perioperative SOX group (Experimental): Participants will receive intravenous cadonilimab (10 mg/kg) in combination with the SOX regimen (oxaliplatin 130 mg/m² and S-1 at a dose of 40-60 mg/m²) for a total of three or four cycles. Subsequently, patients will undergo radical surgery with D2 or D2+ lymphadenectomy. Adjuvant chemotherapy will commence on the 21st or 42st day after surgery, consisting of four cycles of SOX chemotherapy in both groups, administered once every three weeks.
  Interventions: Drug: Neoadjuvant cadonilimab combined with perioperative SOX
- Neoadjuvant placebo plus perioperative SOX (Placebo Comparator): Participants will receive intravenous placebo in combination with the SOX regimen (oxaliplatin 130 mg/m² and S-1 at a dose of 40-60 mg/m²) for a total of three or four cycles. Subsequently, patients will undergo radical surgery with D2 or D2+ lymphadenectomy. Adjuvant chemotherapy will commence on the 21st or 42st day after surgery, consisting of four cycles of SOX chemotherapy in both groups, administered once every three weeks.
  Interventions: Drug: Neoadjuvant placebo plus perioperative SOX

INTERVENTIONS:
Drug: Neoadjuvant cadonilimab combined with perioperative SOX — Cadonilimab: 10 mg/kg, iv, day 1 of every 3 weeks Oxaliplatin: 130 mg/m², iv, day 1 of every 3 weeks S1: 40-60 mg/m², po, day 1-14 of every 3 weeks (BSA < 1.25 m², 40 mg * 2/day, 1.25 m² ≤ BSA < 1.5 m², 50 mg * 2/day, BSA ≥ 1.5 m², 60 mg * 2/day)
  Arms: Neoadjuvant cadonilimab combined with perioperative SOX group
Drug: Neoadjuvant placebo plus perioperative SOX — Placebo: iv, day 1 of every 3 weeks Oxaliplatin: 130 mg/m², iv, day 1 of every 3 weeks S1: 40-60 mg/m², po, day 1-14 of every 3 weeks (BSA < 1.25 m², 40 mg * 2/day, 1.25 m² ≤ BSA < 1.5 m², 50 mg * 2/day, BSA ≥ 1.5 m², 60 mg * 2/day)
  Arms: Neoadjuvant placebo plus perioperative SOX

SUMMARY:
This study aims to investigate the efficacy and safety of neoadjuvant cadonilimab in combination with perioperative SOX chemotherapy, compared to perioperative SOX chemotherapy alone, in patients with diffuse or mixed-type locally advanced gastric or gastroesophageal junction adenocarcinoma. The main questions it seeks to answer are:

1. Is neoadjuvant cadonilimab plus SOX chemotherapy superior to neoadjuvant placebo plus SOX chemotherapy in terms of the pathological complete response (pCR) rate at the time of surgery?
2. To evaluate and compare the 3-year OS rate in patients receiving neoadjuvant cadonilimab plus SOX chemotherapy versus patients receiving placebo plus neoadjuvant SOX chemotherapy regimen.

Participants will be divided into two groups:

1. Experimental group: Participants will receive intravenous cadonilimab (10 mg/kg) in combination with the SOX regimen (oxaliplatin 130 mg/m² and S-1, with the initial dose determined based on body surface area).
2. Control group: Participants will receive a placebo in combination with the SOX regimen.

After completing 3-4 cycles of treatment, patients in both the experimental and control groups will undergo radical surgery with D2 or D2+ lymphadenectomy. Following surgery, patients will receive 4 cycles of adjuvant SOX chemotherapy at 70% of the standard dosage, administered every 21 days, starting within 3-6 weeks post-surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Type of Participant and Disease Characteristics

   1. Patients must have a pathologically confirmed diagnosis of HER-2 negative tumor and diffuse or mixed type gastric or gastroesophageal junction adenocarcinoma according to Lauren's histological subtypes.
   2. Patients must have previously untreated locally advanced gastric or gastroesophageal junction adenocarcinoma (stage cT2, cT3, cT4), with lymph nodes ranging from N1 to N3 and no evidence of metastatic disease (M0).
   3. Patients with Siewert type 2 or 3 tumors are eligible. Enrollment of participants with Siewert type 1 tumors will be limited to those for whom the planned treatment is perioperative chemotherapy and resection.
2. Demographics

   1. Male or female subjects must be between the ages of ≥ 18 and ≤ 75 years at the time of signing the informed consent.
   2. Expected Survival: The expected survival time must be ≥ 12 weeks.
   3. Performance Status: Subjects must have an ECOG performance status of 0 or 1 (refer to Appendix 1).
   4. Male Contraception: Non-sterilized male subjects who are sexually active with a female partner of childbearing potential must use an effective method of contraception from Day 1 through 120 days after receipt of the final dose of the investigational product. It is strongly recommended for the female partner of a male subject to also use an effective method of contraception throughout this period.
   5. Female subjects of childbearing potential must be willing to use adequate contraception methods throughout the study and for 120 days after the last dose of the study drug. The decision to discontinue contraception after this time point should be discussed with the attending physician. Periodic abstinence, contraceptive rhythm methods, and withdrawal are not acceptable forms of contraception.

      * Females of childbearing potential are defined as those who are not surgically sterile (e.g., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).
      * Highly effective contraception methods, resulting in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, are required. Acceptable methods include a combination of a hormonal method (e.g., contraceptive pill) and a barrier method (e.g., male condom plus spermicide) to prevent pregnancy.
      * Barrier methods include male condom plus spermicide, copper T intrauterine device, and levonorgestrel-releasing intrauterine system.
      * Hormonal methods include implants, hormone injection, combined pill, minipill, and patch.
      * If a female subject becomes pregnant or suspects pregnancy during her participation in the study or her partner's participation, she must promptly inform her treating physician.
3. Organ Function

   1. Blood Routine (no blood transfusion within 14 days): WBC ≥ 3.0 × 10^9/L; ANC ≥ 1.5 × 10^9/L; PLT ≥ 100 × 10^9/L; HGB ≥ 80 g/L.
   2. Hepatic Function: Total bilirubin (TBIL) ≤ 1.5 × ULN, or direct bilirubin ≤ ULN for those with total bilirubin levels 1.5 × ULN and ALT/AST levels ≤ 2.5 × ULN.
   3. Renal Function: Creatinine (Cr) ≤ 1.5 × ULN or Creatinine Clearance (CrCl) ≥ 60 mL/min for those with Cr > 1.5 × ULN.
   4. Coagulation Function: INR ≤ 1.5 × ULN, APTT ≤ 1.5 × ULN.
   5. Cardiac Function: Cardiac function will be assessed using electrocardiogram and color Doppler ultrasound, and subjects must have had no myocardial infarction within the last six months. Hypertension and other coronary heart diseases must be controllable.

      * Females of childbearing potential are defined as those who are not surgically sterile (e.g., bilateral tubal ligation, bilateral oophorectomy, or complete hysterectomy) or postmenopausal (defined as 12 months with no menses without an alternative medical cause).
      * Highly effective contraception methods, resulting in a low failure rate (i.e., less than 1% per year) when used consistently and correctly, are required. Acceptable methods include a combination of a hormonal method (e.g., contraceptive pill) and a barrier method (e.g., male condom plus spermicide) to prevent pregnancy.
      * Barrier methods include male condom plus spermicide, copper T intrauterine device, and levonorgestrel-releasing intrauterine system.
      * Hormonal methods include implants, hormone injection, combined pill, minipill, and patch.
      * If a female subject becomes pregnant or suspects pregnancy during her participation in the study or her partner's participation, she must promptly inform her treating physician.
4. Informed Consent All subjects must provide written informed consent to participate in the study.
5. Other Inclusions

   1. Prior Treatment: Patients must not have previously received any anti-tumor treatments, including radiotherapy, chemotherapy, targeted therapy, or immunotherapy.
   2. Plan to proceed to surgery following pre-operative chemotherapy based on standard staging studies per local practice.
   3. Be willing to provide tissue and blood sample from a tumor lesion at baseline and at time of surgery

Exclusion Criteria:

1. Medical Conditions

   1. Has a history of (non-infectious) pneumonitis that required steroids or has current pneumonitis.
   2. Has a known additional malignancy that is progressing or has required active treatment within the past 5 years (except for cutaneous basal cell carcinoma, cutaneous squamous cell carcinoma, or carcinoma in situ that has undergone potentially curative therapy).
   3. Has an active infection requiring systemic therapy.
   4. Has an active autoimmune disease that has required systemic treatment in the past 2 years. (NOTE: Subjects with vitiligo, alopecia, Grave's disease, Type I diabetes mellitus, hypothyroidism (e.g., following Hashimoto's syndrome) only requiring hormone replacement on a stable dose (without adjustment in the first 4 weeks of study treatment), psoriasis or eczema not requiring systemic treatment (within the past 2 years), or conditions not expected to recur in the absence of an external trigger are not excluded.)
   5. Has any complications requiring systemic treatment with corticosteroids such as prednisone (> 10mg/day) or other immunosuppressive medications within 14 days prior to the first administration. Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is allowed.
   6. History of primary immunodeficiency.
   7. Has received a live vaccine or other immune-activating anti-tumor drugs (such as interferon, interleukin, thymosin, or immunotherapy) within 30 days prior to the first dose of study treatment.
   8. Has a known history of active tuberculosis.

      * Known history of allogeneic organ transplantation and allogeneic hematopoietic stem cell transplantation.
   9. Has a known severe allergy or hypersensitivity to cadonilimab or sintilimab or any of the study chemotherapy agents and/or to any of their excipients.
   10. Presence of any of the following cardiovascular and cerebrovascular diseases or cardiovascular and cerebrovascular risk factors:

       * Grade II or higher myocardial ischemia or myocardial infarction, poorly controlled arrhythmia (including QTc interval ≥ 480 ms), grade III or IV cardiac insufficiency, or left ventricular ejection fraction (LVEF) < 50.0% as determined by color Doppler echocardiography.
       * Cerebrovascular accident, transient ischemic attack, or other arteriovenous thrombotic, embolic, or ischemic events.
2. Prior/Concomitant Therapy

   1. Subjects who have already enrolled in another clinical study, unless it is an observational, non-interventional clinical study, or they are in the follow-up period for an interventional study (the time between the first dose of cadonilimab and the last dose in the previous clinical study should be more than 4 weeks or 5 times the half-life of the previous study drug).
   2. Subjects who have received any systemic or curative anti-tumor therapy, including radiotherapy, chemotherapy, targeted therapy.
   3. Subjects who have previously received any anti-PD-1, anti-PD-L1, anti-CTLA-4 antibody, or any other antibody or drug therapy targeting T-cell co-stimulation or checkpoint pathway, e.g. ICOS or agonists (e.g., CD40, CD137, GITR, and OX40, etc.).
3. Other exclusion criteria

   1. Confirmed HER-2 positive tumor will be excluded.
   2. Patients could not provide tumor samples and blood samples.
   3. Pregnant or lactating patients, as well as patients with childbearing potential who plan to be pregnant within 5 months after the study; Women of childbearing should receive a blood pregnancy test within 7 days before the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 668 (Estimated)
Dates: Start 2025-05-15 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Pathological complete response (pCR) rate | From enrollment to surgical treatment, it is expected to require 4 months.
  The pCR is defined as no invasive disease within an entirely submitted and evaluated gross lesion, and histologically negative nodes as assessed by BIPR based on Becker regression criteria. pCR rate is defined as the proportion of participants having pCR.
3-year survival rate (3-year OS rate) | 3 years
  3-year OS rate is defined as the proportion of patients alive at 3 years after randomization estimated using the Kaplan-Meier method. Participants without documented death at the time of analysis will be censored at the date of last known alive.

SECONDARY OUTCOMES:
Major pathological response (MPR) rate | From enrollment to surgical treatment, it is expected to require 4 months.
  MPR rate by BIPR is defined as the proportion of patients with ≤ 10% residual viable tumor in the resected primary tumor and all resected lymph nodes after completion of neoadjuvant therapy as assessed by BIPR.
Objective response rate (ORR) | From enrollment to preoperative imaging evaluation, it is expected to require 3-4 months.
  ORR is defined as the proportion of patients who had complete response (CR) or partial response (PR) as assessed by BICR per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST v1.1) in all randomized patients with measurable disease at baseline.
Treatment emergent adverse event | From enrollment to the completion or discontinuation of treatment, an estimated duration of eight months is expected.
  Incidence and severity of TEAEs, including serious adverse events (SAEs) and immune-mediated adverse events (imAEs), with severity determined according to National Cancer Institute-Common Terminology Criteria for Adverse Events Version 5.0 (NCI-CTCAE v5.0).
Disease control rate (DCR) | From enrollment to preoperative imaging evaluation, it is expected to require 3-4 months.
  DCR is defined as the proportion of patients who had CR, PR or stable disease (SD) as assessed by BICR per RECIST v1.1 in all randomized patients with measurable disease at baseline.
3-year BICR-assessed disease-free survival (DFS) rate | 3 years
  3-year BICR-assessed DFS rate is defined as the time from the first date of surgery with R0 resection to local or distant recurrence or death due to any cause, whichever occurs first, as determined by BICR during the adjuvant treatment and safety follow-up.
R0 resection rate | From enrollment to surgical treatment, it is expected to require 4 months.
  R0 resection rate is defined as the proportion of patients who had no cancer cells could be found at the surgical margins under the microscope, indicating complete removal of the lesion with no residual tumor visible either macroscopically or microscopically.
Surgery-related complications | After the completion of surgery, it is expected to take 5 months.
  Surgery-related complications is defined as patients who received surgery within 30 days and experienced any grade surgery-related complications per Clavien-Dindo Classification of Surgical Complications, including vomiting, fever, incision infection, post-operative pneumonia, anastomotic hemorrhage or leakage, chylous leakage, pneumonia, intestinal obstruction, etc,
Tumor downstage rate | After the completion of surgery, it is expected to take 4 months.
  The tumor downstage rate is defined as the proportion of patients who had overall ypTNM or T or N stage was decreased from cTNM, cT or cN stage at baseline. Tumor stage was evaluated based on baseline cTNM stage and postoperative ypTNM stage according to the 8th edition of the AJCC Gastric Cancer Stage.
Programmed death ligand-1 Combined Positive Score (PD-L1 CPS) | Baseline
  PD-L1 expression as the predictive biomarker for efficacy (including but not limited to pCR rate, MPR rate, 3-year OS rate, and 3-year DFS rate). The CPS score ranges from 0 to 100. High levels of PD-L1 expression are usually associated with better responses to immunotherapy, and patients may benefit more from immune checkpoint inhibitors.
Microsatellite Instability (MSI) | Baseline
  The status of MSI as the predictive biomarker for efficacy (including but not limited to pCR rate, MPR rate, 3-year OS rate, and 3-year DFS rate).

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Gansu Provincial Hospital, Lanzhou, Gansu
  - Lanzhou University Second Hospital, Lanzhou, Gansu
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - The Gastrointestinal Surgery Department, Sun Yat-sen University Cancer Center Gansu Hospital, Lanzhou, Gansu

IPD SHARING:
Plan to Share IPD: No